CLINICAL TRIAL: NCT04004312
Title: Single Fractions SBRT in the Treatment of Prostate Cancer: A Phase I Study
Brief Title: Single Fractions SBRT for Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fabio Cury (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Fabio Cury, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-4650
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: single fraction; SBRT; Space OAR Gel
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Fraction SBRT in the treatment of prostate cancer (Experimental): Prior to treatment, a hydrogel spacer will be inserted between the recutm and prostate. A urinary catheter will also be inserted in the bladder. A single dose of 19Gy will be delivered with an IMRT technique. The treatment should last approximately 30 minutes. After the treatment, the urinary catheter will be removed.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Shorter radiation therapy means that a higher dose will be offered. To limit side effects of exposure to a high dose, a medical device protecting the rectum will be used. The medical device to be used is called SpaceOAR hydrogel (device). The SpaceOAR hydrogel creates space between the rectum and the prostate, making it much less likely that the rectum is exposed to radiation. It is injected into place prior to the start of radiation treatment using a needle. Patients may be awake or asleep under local anesthesia for the procedure. SpaceOAR hydrogel is not painful, it remains stable during radiation therapy and then is gradually absorbed by the body over the course of approximately six months, once radiation therapy has been completed.
  Other Names: Space OAR Gel

SUMMARY:
It is a phase I study of radical hypofractionation delivering one single fraction of SBRT in patients with low- and favorable intermediate-risk prostate cancer that will undergo placement of the SpaceOAR hydrogel prior to treatment.

Our hypothesis is that treatments can be safely delivered in one single fraction using SBRT provided the separation between the prostate and rectum is increased using the hydrogel

DETAILED DESCRIPTION:
There is a pre-treatment visit to the radiation oncology department. A gel is injected between the prostate and the rectum. This procedure is done with the use of a transrectal ultrasound, similarly to the prostate biopsy the patient had. A local anesthetic will be applied to numb the skin and to the underneath tissue where the injection will be performed. The procedure itself will take approximately 20 minutes and after a short observation time, the patient returns home.

The next visit (approximately after 7 days after the insertion of the gel), a CT scan and MRI-scan will be done. Prior to the scans, a urinary catheter will be inserted in the bladder through the penis, and removed once the scans are done. Using these images, the doctor and the team involved will perform an individualized planning study to establish the safest way the radiation will enter your body. When the treatment plan is ready, patient is called to receive the single treatment.

A urinary catheter again will be inserted in the bladder and the patient will be directed to the room where your treatment will be delivered. The treatment should last approximately 30 minutes. After the treatment, the urinary catheter will be removed.

ELIGIBILITY:
Inclusion Criteria:

Histologically proven adenocarcinoma of the prostate. Tl-2b (AJCC 7th edition) Gleason score 6 or 7 (3+4)) or Gleason 7(4+3) and recent PSA < 10 (less than 30 days; must obtained >90 days from stopping dutasteride or >30 days from stopping finasteride)

Recent PSA under 15 ng/dL (less than 30 days; must obtained >90 days from stopping dutasteride or >30 days from stopping finasteride) OR Gleason 7(4+3) and recent PSA < 10 (less than 30 days; must obtained >90 days from stopping dutasteride or >30 days from stopping finasteride)

International Prostate Symptom Score <16 Prostate gland volume< 80cc

Zubrod Performance Status 0-1 within 60 days prior to registration

Age >: 18

Patient must be able to provide study-specific informed consent prior to study entry.

Exclusion Criteria:

Patients who opt to receive another treatment modality, such as surgery, or undergo active surveillance.

Prior or concurrent invasive malignancy (except non-melanomatous skin cancer) or lymphomatous/hematogenous malignancy unless continually disease free for a minimum of 5 years. All patients with in situ carcinoma are eligible for this study (for example, carcinoma in situ of the oral cavity) except patients with carcinoma of the bladder (including in situ bladder cancer or superficial bladder cancer).

Evidence of distant metastases

Regional lymph node involvement

Previous radical surgery (prostatectomy), cryosurgery, or HIFU for prostate cancer Previous pelvic irradiation, prostate brachytherapy, or bilateral orchiectomy Previous hormonal therapy, such as LHRH agonists or antagonists, anti-androgens, estrogens, or surgical castration (orchiectomy)

Use of finasteride within 30 days prior to registration. PSA should not be obtained prior to 30 days after stopping finasteride.

Use of dutasteride within 90 days prior to registration. PSA should not be obtained prior to 90 days after stopping dutasteride.

Previous or concurrent cytotoxic chemotherapy for prostate cancer Severe, active co-morbidity, defined as follows:

Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months

Transmural myocardial infarction within the last 6 months

Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration

Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration

Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol. (Patients on Coumadin or other blood thinning agents are eligible for this study.)

Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Estimated)
Dates: Start 2018-11-07 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Small bowel or rectal irritation, | 3 months
  To assess acute gastro-intestinal (GI) toxicity such as abdominal cramping, diarrhea, rectal urgency, proctitis, or hematochezia;
Bladder complications | 3 months
  Bladder complications including urinary frequency/urgency, dysuria, hematuria, urinary tract infection, and incontinence;

SECONDARY OUTCOMES:
To assess late GI and GU toxicity | 3 years
  gastro-intestinal (GI) toxicity such as abdominal cramping, diarrhea, rectal urgency, proctitis, or hematochezia;and GU toxicity such as Bladder complications including urinary frequency/urgency, dysuria, hematuria, urinary tract infection, and incontinence;
PSA control | 5 years
  To assess the rate of biochemical control

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Cury, MD, Principal Investigator — McGill University Health Centre- Cedars Cancer Centre
Locations (1):
- McGill University Health Centre-Cedars Cancer Centre, Montreal, Quebec, Canada

REFERENCES:
- [Background] King CR, Fowler JF. A simple analytic derivation suggests that prostate cancer alpha/beta ratio is low. Int J Radiat Oncol Biol Phys. 2001 Sep 1;51(1):213-4. doi: 10.1016/s0360-3016(01)01651-0. No abstract available. PMID 11516871
- [Background] Fowler JF, Ritter MA, Chappell RJ, Brenner DJ. What hypofractionated protocols should be tested for prostate cancer? Int J Radiat Oncol Biol Phys. 2003 Jul 15;56(4):1093-104. doi: 10.1016/s0360-3016(03)00132-9. PMID 12829147
- [Background] King CR, Brooks JD, Gill H, Presti JC Jr. Long-term outcomes from a prospective trial of stereotactic body radiotherapy for low-risk prostate cancer. Int J Radiat Oncol Biol Phys. 2012 Feb 1;82(2):877-82. doi: 10.1016/j.ijrobp.2010.11.054. Epub 2011 Feb 6. PMID 21300474
- [Background] Katz AJ, Santoro M, Ashley R, Diblasio F, Witten M. Stereotactic body radiotherapy for organ-confined prostate cancer. BMC Urol. 2010 Feb 1;10:1. doi: 10.1186/1471-2490-10-1. PMID 20122161
- [Background] Fuller DB, Naitoh J, Lee C, Hardy S, Jin H. Virtual HDR CyberKnife treatment for localized prostatic carcinoma: dosimetry comparison with HDR brachytherapy and preliminary clinical observations. Int J Radiat Oncol Biol Phys. 2008 Apr 1;70(5):1588-97. doi: 10.1016/j.ijrobp.2007.11.067. PMID 18374232
- [Background] Faria S, Ruo R, Cury F, Duclos M, Souhami L. Acute and late toxicity in high-risk prostate cancer patients treated with androgen suppression and hypofractionated pelvic radiation therapy. Pract Radiat Oncol. 2017 Jul-Aug;7(4):264-269. doi: 10.1016/j.prro.2017.01.003. Epub 2017 Jan 20. PMID 28222995
- [Background] Faria SL, Neto OB, Cury F, Shenouda G, Russel R, Souhami L. Moderate hypofractionated external beam radiotherapy alone for intermediate risk prostate cancer: long term outcomes. Can J Urol. 2016 Apr;23(2):8209-14. PMID 27085825
- [Background] Patel N, Faria S, Cury F, David M, Duclos M, Shenouda G, Ruo R, Souhami L. Hypofractionated radiation therapy (66 Gy in 22 fractions at 3 Gy per fraction) for favorable-risk prostate cancer: long-term outcomes. Int J Radiat Oncol Biol Phys. 2013 Jul 1;86(3):534-9. doi: 10.1016/j.ijrobp.2013.02.010. Epub 2013 Apr 15. PMID 23597418
- [Background] Rene N, Faria S, Cury F, David M, Duclos M, Shenouda G, Souhami L. Hypofractionated radiotherapy for favorable risk prostate cancer. Int J Radiat Oncol Biol Phys. 2010 Jul 1;77(3):805-10. doi: 10.1016/j.ijrobp.2009.05.047. PMID 20510194
- [Background] Catton CN, Lukka H, Gu CS, Martin JM, Supiot S, Chung PWM, Bauman GS, Bahary JP, Ahmed S, Cheung P, Tai KH, Wu JS, Parliament MB, Tsakiridis T, Corbett TB, Tang C, Dayes IS, Warde P, Craig TK, Julian JA, Levine MN. Randomized Trial of a Hypofractionated Radiation Regimen for the Treatment of Localized Prostate Cancer. J Clin Oncol. 2017 Jun 10;35(17):1884-1890. doi: 10.1200/JCO.2016.71.7397. Epub 2017 Mar 15. PMID 28296582
- [Background] Lee WR, Dignam JJ, Amin MB, Bruner DW, Low D, Swanson GP, Shah AB, D'Souza DP, Michalski JM, Dayes IS, Seaward SA, Hall WA, Nguyen PL, Pisansky TM, Faria SL, Chen Y, Koontz BF, Paulus R, Sandler HM. Randomized Phase III Noninferiority Study Comparing Two Radiotherapy Fractionation Schedules in Patients With Low-Risk Prostate Cancer. J Clin Oncol. 2016 Jul 10;34(20):2325-32. doi: 10.1200/JCO.2016.67.0448. Epub 2016 Apr 4. PMID 27044935
- [Background] Dearnaley D, Syndikus I, Mossop H, Khoo V, Birtle A, Bloomfield D, Graham J, Kirkbride P, Logue J, Malik Z, Money-Kyrle J, O'Sullivan JM, Panades M, Parker C, Patterson H, Scrase C, Staffurth J, Stockdale A, Tremlett J, Bidmead M, Mayles H, Naismith O, South C, Gao A, Cruickshank C, Hassan S, Pugh J, Griffin C, Hall E; CHHiP Investigators. Conventional versus hypofractionated high-dose intensity-modulated radiotherapy for prostate cancer: 5-year outcomes of the randomised, non-inferiority, phase 3 CHHiP trial. Lancet Oncol. 2016 Aug;17(8):1047-1060. doi: 10.1016/S1470-2045(16)30102-4. Epub 2016 Jun 20. PMID 27339115
- [Background] Tang CI, Loblaw DA, Cheung P, Holden L, Morton G, Basran PS, Tirona R, Cardoso M, Pang G, Gardner S, Cesta A. Phase I/II study of a five-fraction hypofractionated accelerated radiotherapy treatment for low-risk localised prostate cancer: early results of pHART3. Clin Oncol (R Coll Radiol). 2008 Dec;20(10):729-37. doi: 10.1016/j.clon.2008.08.006. Epub 2008 Oct 5. PMID 18838256
- [Background] McBride SM, Wong DS, Dombrowski JJ, Harkins B, Tapella P, Hanscom HN, Collins SP, Kaplan ID. Hypofractionated stereotactic body radiotherapy in low-risk prostate adenocarcinoma: preliminary results of a multi-institutional phase 1 feasibility trial. Cancer. 2012 Aug 1;118(15):3681-90. doi: 10.1002/cncr.26699. Epub 2011 Dec 13. PMID 22170628
- [Background] Madsen BL, Hsi RA, Pham HT, Fowler JF, Esagui L, Corman J. Stereotactic hypofractionated accurate radiotherapy of the prostate (SHARP), 33.5 Gy in five fractions for localized disease: first clinical trial results. Int J Radiat Oncol Biol Phys. 2007 Mar 15;67(4):1099-105. doi: 10.1016/j.ijrobp.2006.10.050. PMID 17336216
- [Background] Loblaw A, Cheung P, D'Alimonte L, Deabreu A, Mamedov A, Zhang L, Tang C, Quon H, Jain S, Pang G, Nam R. Prostate stereotactic ablative body radiotherapy using a standard linear accelerator: toxicity, biochemical, and pathological outcomes. Radiother Oncol. 2013 May;107(2):153-8. doi: 10.1016/j.radonc.2013.03.022. Epub 2013 May 3. PMID 23647750
- [Background] Lin YW, Lin LC, Lin KL. The early result of whole pelvic radiotherapy and stereotactic body radiotherapy boost for high-risk localized prostate cancer. Front Oncol. 2014 Oct 31;4:278. doi: 10.3389/fonc.2014.00278. eCollection 2014. PMID 25401085
- [Background] Ju AW, Wang H, Oermann EK, Sherer BA, Uhm S, Chen VJ, Pendharkar AV, Hanscom HN, Kim JS, Lei S, Suy S, Lynch JH, Dritschilo A, Collins SP. Hypofractionated stereotactic body radiation therapy as monotherapy for intermediate-risk prostate cancer. Radiat Oncol. 2013 Jan 31;8:30. doi: 10.1186/1748-717X-8-30. PMID 23369294
- [Background] King CR, Freeman D, Kaplan I, Fuller D, Bolzicco G, Collins S, Meier R, Wang J, Kupelian P, Steinberg M, Katz A. Stereotactic body radiotherapy for localized prostate cancer: pooled analysis from a multi-institutional consortium of prospective phase II trials. Radiother Oncol. 2013 Nov;109(2):217-21. doi: 10.1016/j.radonc.2013.08.030. Epub 2013 Sep 20. PMID 24060175
- [Background] Friedland JL, Freeman DE, Masterson-McGary ME, Spellberg DM. Stereotactic body radiotherapy: an emerging treatment approach for localized prostate cancer. Technol Cancer Res Treat. 2009 Oct;8(5):387-92. doi: 10.1177/153303460900800509. PMID 19754215
- [Background] Chen LN, Suy S, Uhm S, Oermann EK, Ju AW, Chen V, Hanscom HN, Laing S, Kim JS, Lei S, Batipps GP, Kowalczyk K, Bandi G, Pahira J, McGeagh KG, Collins BT, Krishnan P, Dawson NA, Taylor KL, Dritschilo A, Lynch JH, Collins SP. Stereotactic body radiation therapy (SBRT) for clinically localized prostate cancer: the Georgetown University experience. Radiat Oncol. 2013 Mar 13;8:58. doi: 10.1186/1748-717X-8-58. PMID 23497695
- [Background] Bolzicco G, Favretto MS, Scremin E, Tambone C, Tasca A, Guglielmi R. Image-guided stereotactic body radiation therapy for clinically localized prostate cancer: preliminary clinical results. Technol Cancer Res Treat. 2010 Oct;9(5):473-7. doi: 10.1177/153303461000900505. PMID 20815418
- [Background] Katz AJ, Kang J. Stereotactic body radiotherapy as treatment for organ confined low- and intermediate-risk prostate carcinoma, a 7-year study. Front Oncol. 2014 Sep 2;4:240. doi: 10.3389/fonc.2014.00240. eCollection 2014. PMID 25229051
- [Background] Davis J, Sharma S, Shumway R, Perry D, Bydder S, Simpson CK, D'Ambrosio D. Stereotactic Body Radiotherapy for Clinically Localized Prostate Cancer: Toxicity and Biochemical Disease-Free Outcomes from a Multi-Institutional Patient Registry. Cureus. 2015 Dec 4;7(12):e395. doi: 10.7759/cureus.395. PMID 26798571
- [Background] Katz A, Formenti SC, Kang J. Predicting Biochemical Disease-Free Survival after Prostate Stereotactic Body Radiotherapy: Risk-Stratification and Patterns of Failure. Front Oncol. 2016 Jul 8;6:168. doi: 10.3389/fonc.2016.00168. eCollection 2016. PMID 27458572
- [Background] Kim DN, Straka C, Cho LC, Lotan Y, Yan J, Kavanagh B, Raben D, Cooley S, Brindle J, Xie XJ, Pistenmaa D, Timmerman R. Early and multiple PSA bounces can occur following high-dose prostate stereotactic body radiation therapy: Subset analysis of a phase 1/2 trial. Pract Radiat Oncol. 2017 Jan-Feb;7(1):e43-e49. doi: 10.1016/j.prro.2016.06.010. Epub 2016 Jun 24. PMID 27637137
- [Background] Quon HC, Musunuru HB, Cheung P, Pang G, Mamedov A, D'Alimonte L, Deabreu A, Zhang L, Loblaw A. Dose-Escalated Stereotactic Body Radiation Therapy for Prostate Cancer: Quality-of-Life Comparison of Two Prospective Trials. Front Oncol. 2016 Aug 29;6:185. doi: 10.3389/fonc.2016.00185. eCollection 2016. PMID 27622157
- [Background] Avkshtol V, Dong Y, Hayes SB, Hallman MA, Price RA, Sobczak ML, Horwitz EM, Zaorsky NG. A comparison of robotic arm versus gantry linear accelerator stereotactic body radiation therapy for prostate cancer. Res Rep Urol. 2016 Aug 18;8:145-58. doi: 10.2147/RRU.S58262. eCollection 2016. PMID 27574585
- [Background] Prada PJ, Cardenal J, Blanco AG, Anchuelo J, Ferri M, Fernandez G, Arrojo E, Vazquez A, Pacheco M, Fernandez J. High-dose-rate interstitial brachytherapy as monotherapy in one fraction for the treatment of favorable stage prostate cancer: Toxicity and long-term biochemical results. Radiother Oncol. 2016 Jun;119(3):411-6. doi: 10.1016/j.radonc.2016.04.006. Epub 2016 Apr 22. PMID 27118583
- [Background] Jawad MS, Dilworth JT, Gustafson GS, Ye H, Wallace M, Martinez A, Chen PY, Krauss DJ. Outcomes Associated With 3 Treatment Schedules of High-Dose-Rate Brachytherapy Monotherapy for Favorable-Risk Prostate Cancer. Int J Radiat Oncol Biol Phys. 2016 Mar 15;94(4):657-66. doi: 10.1016/j.ijrobp.2015.10.011. Epub 2015 Nov 10. PMID 26797541
- [Background] Hoskin P, Rojas A, Lowe G, Bryant L, Ostler P, Hughes R, Milner J, Cladd H. High-dose-rate brachytherapy alone for localized prostate cancer in patients at moderate or high risk of biochemical recurrence. Int J Radiat Oncol Biol Phys. 2012 Mar 15;82(4):1376-84. doi: 10.1016/j.ijrobp.2011.04.031. Epub 2011 Jun 15. PMID 21680108
- [Background] Ghilezan M, Martinez A, Gustason G, Krauss D, Antonucci JV, Chen P, Fontanesi J, Wallace M, Ye H, Casey A, Sebastian E, Kim L, Limbacher A. High-dose-rate brachytherapy as monotherapy delivered in two fractions within one day for favorable/intermediate-risk prostate cancer: preliminary toxicity data. Int J Radiat Oncol Biol Phys. 2012 Jul 1;83(3):927-32. doi: 10.1016/j.ijrobp.2011.05.001. Epub 2011 Dec 23. PMID 22197086
- [Background] Morton G, Chung HT, McGuffin M, Helou J, D'Alimonte L, Ravi A, Cheung P, Szumacher E, Liu S, Al-Hanaqta M, Zhang L, Mamedov A, Loblaw A. Prostate high dose-rate brachytherapy as monotherapy for low and intermediate risk prostate cancer: Early toxicity and quality-of life results from a randomized phase II clinical trial of one fraction of 19Gy or two fractions of 13.5Gy. Radiother Oncol. 2017 Jan;122(1):87-92. doi: 10.1016/j.radonc.2016.10.019. Epub 2016 Nov 4. PMID 27823821
- [Background] Anwar M, Weinberg V, Seymour Z, Hsu IJ, Roach M 3rd, Gottschalk AR. Outcomes of hypofractionated stereotactic body radiotherapy boost for intermediate and high-risk prostate cancer. Radiat Oncol. 2016 Jan 21;11:8. doi: 10.1186/s13014-016-0585-y. PMID 26792201
- [Background] Hamstra DA, Mariados N, Sylvester J, Shah D, Karsh L, Hudes R, Beyer D, Kurtzman S, Bogart J, Hsi RA, Kos M, Ellis R, Logsdon M, Zimberg S, Forsythe K, Zhang H, Soffen E, Francke P, Mantz C, Rossi P, DeWeese T, Daignault-Newton S, Fischer-Valuck BW, Chundury A, Gay H, Bosch W, Michalski J. Continued Benefit to Rectal Separation for Prostate Radiation Therapy: Final Results of a Phase III Trial. Int J Radiat Oncol Biol Phys. 2017 Apr 1;97(5):976-985. doi: 10.1016/j.ijrobp.2016.12.024. Epub 2016 Dec 23. PMID 28209443